CLINICAL TRIAL: NCT00020449
Title: A Phase II Study of Liposomal Doxorubicin and Interleukin-12 in AIDS-Associated Kaposi's Sarcoma Followed by Chronic Administration of Interleukin-12
Brief Title: Liposomal Doxorubicin and Interleukin-12 in Treating Patients With AIDS-Related Kaposi's Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068502; NCI-01-C-0067; NCI-4010; NCT00008879 (obsolete NCT alias)
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2004-03

CONDITIONS: Sarcoma
Keywords: AIDS-related Kaposi sarcoma; recurrent Kaposi sarcoma
MeSH Terms: conditions — Sarcoma; AIDS-related Kaposi sarcoma; Sarcoma, Kaposi | interventions — Interleukin-12 Subunit p35; Paclitaxel

INTERVENTIONS:
Biological: recombinant interleukin-12
Drug: paclitaxel
Drug: pegylated liposomal doxorubicin hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop tumor cells from dividing so they stop growing or die. Interleukin-12 may kill tumor cells by stopping blood flow to the tumor and by stimulating a person's white blood cells to kill the tumor cells. Combining chemotherapy with interleukin-12 may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining liposomal doxorubicin with interleukin-12 in treating patients who have AIDS-related Kaposi's sarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the overall response rate in patients with AIDS-associated Kaposi's sarcoma (KS) treated with doxorubicin HCl liposome and interleukin-12.
* Determine the time to response and the number of complete responses in patients treated with this regimen.
* Determine the progression-free survival of patients treated with this regimen.
* Provide pilot information on the ability of interleukin-12 to maintain major responses induced with paclitaxel salvage therapy in patients with aggressive or life-threatening KS after treatment failure with doxorubicin HCl liposome and interleukin-12.
* Determine the effect of this regimen on CD4 counts and viral load in these patients.

OUTLINE: Patients receive doxorubicin HCl liposome (LipoDox) IV over 30 minutes once every 3 weeks for a total of 6 doses. Beginning concurrently with the initiation of LipoDox, patients also receive interleukin-12 (IL-12) subcutaneously twice weekly (at least 3 days apart) for up to 3 years.

Patients with refractory disease are transferred to the paclitaxel salvage therapy regimen comprising paclitaxel IV continuously on days 1-4 once every 3 weeks until a major response is achieved. Beginning concurrently with the initiation of paclitaxel salvage therapy, patients also receive IL-12 as above for up to 3 years.

Treatment continues in the absence of disease progression or unacceptable toxicity. Patients achieving a complete response may discontinue IL-12 administration. If necessary, IL-12 treatment may resume at a later time.

Patients are followed at 4 weeks.

PROJECTED ACCRUAL: A total of 24-36 patients will be accrued for this study within 2-4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed Kaposi's sarcoma (KS)
* HIV positive
* Evaluable disease involving the skin and/or viscera

  * At least 5 lesions not previously treated with local therapy if restricted to the skin
  * Pulmonary lesions evaluable by CT scan
  * Gastrointestinal lesions evaluable by visualization or fiberoptic instrumentation
* Presence of at least one of the following indications for cytotoxic chemotherapy:

  * Pulmonary involvement
  * Visceral involvement
  * Pain
  * Edema
  * Ulcerating lesions
  * Decreased range of joint motion due to KS
  * Multiple lesions not amenable to local therapy
  * Lymphedema that impairs mobility or range of motion
  * Significant psychological impact leading to social withdrawal
* Progressive disease within the past 3 weeks while receiving a stable regimen of highly active antiretroviral therapy for at least 4 weeks unless there is a need for urgent chemotherapy
* Prior participation on this study allowed, provided patient was removed from study due to non-pancreatic hyperamylasemia and the following are true:

  * No dose-limiting toxicity by clinical and laboratory assessment
  * Pancreatic amylase portion normal by fractionated amylase
  * Lipase normal
  * No symptoms referable to the pancreas

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 30-100%

Life expectancy:

* More than 2 months

Hematopoietic:

* Hemoglobin at least 9.0 g/dL
* Absolute neutrophil count at least 750/mm^3
* Platelet count at least 75,000/mm^3

Hepatic:

* Bilirubin no greater than 3.8 mg/dL with direct fraction no greater than 0.3 mg/dL and indirect fraction no greater than 3.5 mg/dL if due to protease inhibitor therapy
* PT or aPTT no greater than 120% of control unless due to lupus-type anticoagulant
* AST no greater than 2.5 times upper limit of normal
* No prior hepatic cirrhosis
* No hepatic dysfunction

Renal:

* Creatinine no greater than 1.5 mg/dL
* Creatinine clearance at least 60 mL/min

Cardiovascular:

* No congestive heart failure
* Ejection fraction at least 40% by MUGA or echocardiogram

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception during and for 2 months after study participation
* No clinically significant autoimmune disease
* No active, gross gastrointestinal bleeding or uncontrolled peptic ulcer disease
* No prior inflammatory bowel disease
* No other prior or concurrent malignancy except squamous cell carcinoma in situ of the cervix or anus, completely resected basal cell carcinoma, or malignancy in complete remission for at least 1 year from the time a response was first documented
* No severe or life-threatening infection within the past 2 weeks
* No abnormality that would be scored as grade 3 toxicity except lymphopenia or direct manifestations of KS
* No known hypersensitivity to interleukin-12 (IL-12) or other compounds known to cross-react with IL-12
* No other medical condition that would preclude study entry

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* More than 2 weeks since prior cytokines or colony-stimulating factors other than epoetin alfa, filgrastim (G-CSF), or sargramostim (GM-CSF)
* No prior combination interleukin-12 and doxorubicin HCl liposome except for patients previously treated on this protocol who are being enrolled for paclitaxel salvage therapy
* No concurrent immunomodulatory agents
* No concurrent cytokines except epoetin alfa or G-CSF

Chemotherapy:

* See Disease Characteristics
* See Biologic therapy
* At least 3 weeks since prior chemotherapy (6 weeks for mitomycin or nitrosoureas)
* More 6 months since prior suramin
* No other concurrent cytotoxic chemotherapy

Endocrine therapy:

* More than 2 months since prior systemic glucocorticoid steroids at doses sufficient to affect immune response (e.g., more than 20 mg of prednisone for more than 1 week)
* Concurrent replacement glucocorticoid therapy allowed
* No other concurrent systemic glucocorticoid therapy

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* Concurrent antiretroviral therapy required
* No other concurrent anti-KS therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-01; Study Completion 2004-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pallavi P. Kumar, MD, Study Chair — NCI - HIV and AIDS Malignancy Branch
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland, United States

REFERENCES:
- [Result] Little RF, Aleman K, Kumar P, Wyvill KM, Pluda JM, Read-Connole E, Wang V, Pittaluga S, Catanzaro AT, Steinberg SM, Yarchoan R. Phase 2 study of pegylated liposomal doxorubicin in combination with interleukin-12 for AIDS-related Kaposi sarcoma. Blood. 2007 Dec 15;110(13):4165-71. doi: 10.1182/blood-2007-06-097568. Epub 2007 Sep 10. PMID 17846226
- [Result] Little RF, Aleman K, Merced K, et al.: Preliminary results of combination liposomal doxorubicin and interleukin-12 followed by chronic IL-12 maintenance therapy in advanced AIDS-related Kaposi's sarcoma. [Abstract] 10th Conference on Retroviruses and Opportunistic Infections, February 10-14, 2003, Boston, Massachusetts A-816, 2003.